CLINICAL TRIAL: NCT02987439
Title: COPD-EXA-REHAB. Early Pulmonary Rehabilitation of Patients With Acute Exacerbation of COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Jon Torgny Wilcke, Associate Professor, Pricipal Investigator, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-2-2013-143
Record Dates: First submitted 2016-12-06; First posted 2016-12-09 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Chronic Obstructive Lung Disease
Keywords: COPD; Exacerbation; Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard care group (No Intervention): * Standard medical treatment for the exacerbation of COPD
  * Standard medical treatment of COPD according to GOLD
  * A visit by a pulmonary nurse at the patients own home 3-5 days after discharge. Lung function and smoking history is recorded. Correct use of inhaler is instructed.
  * Visit in the outpatient clinic within the next 2-6 months after discharge as follow-up
  * In the outpatient clinic they will receive an offer of pulmonary rehabilitation
- Rehabilitation group (Experimental): The group will begin pulmonary rehabilitation during hospital admission. Afterwards a rehabilitation program twice weekly for 7 weeks.
  Beside rehabilitation they will receive same treatment as the standard care group
  Interventions: Other: Pulmonary rehabilitation

INTERVENTIONS:
Other: Pulmonary rehabilitation — The intervention is pulmonary rehabilitation
  Arms: Rehabilitation group

SUMMARY:
Purpose: In a randomized controlled trial we will assess the effect of early pulmonary rehabilitation in patient with an acute exacerbation of chronic obstructive lung disease (AECOPD).

DETAILED DESCRIPTION:
Background:

Pulmonary rehabilitation is a key element in treatment of stable COPD. A Cochrane review from 2011 showed that early pulmonary rehabilitation for COPD exacerbation 6-10 days after discharge, or during prolonged hospitalization significantly reduced mortality and hospitalizations without serious side effects. It consist of 9 small studies and larger RCT studies is required to establish the effect of early pulmonary rehabilitation.

AIM: The aim of the study is to investigate whether early pulmonary rehabilitation can reduce mortality og hospitalization in patients with acute exacerbation of COPD. Secondary increase exercise capacity, reduce symptoms and improve quality of life.

Methods:

Design: The study is a single center randomized, controlled, open label trial, with an intervention group and a control group. The patients are randomized to either a prespecified rehabilitation program, which is standardized to patients with COPD, or usual care. The patients' data are being recorded at baseline and visits at 2 and 6 months: Lung function (FEV1, FVC), CO in exhaled air, O2 saturation in the blood (and possibly O2 supplement), Heart Rate, Dyspnoea (Borg scale and Medical Research Council (MRC scale)), Quality of life (CAT), Walk Test (ISWT and ESWT), Daily medication, Outdoor activity. Information on mortality, hospital admissions, emergency room visits after 6 and 12 months is obtained from relevant databases.

Population: Patients Hospitalized with an exacerbation of COPD to the department of respiratory medicine at Gentofte Hospital. The inclusion criteria are: A diagnose of COPD, Age >18, expected discharge to own homes, can walk 10 meters independently (with or without a walking aid). Exclusion criteria are: Life expectancy <6 months due to another illness (cancer, severe heart disease, etc.), difficulties in understanding and speaking Danish (e.g. due to dementia), place of residence outside Gentofte Hospital admission area.

Randomization: A total of 150 COPD patients will be included. The participants are randomized to early rehabilitation or usual care in a 1:1 ratio, using a computer-generated block-randomization for each center. The participant is presented with a sealed envelope containing a piece of paper with either "A" (= REHAB) or "B" (= usual care). The randomization list is stored at Gentofte Hospital in a sealed envelope.

A participant who is readmitted will not be re-randomized.

Patients arre introduced to an acute telephone hotline, operated by a nurse.

The patients in the intervention group will during Hospitalization begin the rehabilitation program. The program consist of exercise training, breathing techniques and education. Before discharge the patients will be assessed to either A: outpatient rehabilitation in hospital or community clinic or B: Rehabilitation in their own homes twice weekly in 7 weeks

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to hospital with acute exacerbation of COPD to Department Respiratory Medicine, Gentofte Hospital
* Verified diagnosis of COPD FEV1/FVC <70 % in stable phase.
* Expected discharge to their own home.
* Minimal of 10 meters walking distance independently
* Oral and written consent
* Age > 18 year

Exclusion Criteria:

* Life expectancy <6 months due to another illness (cancer, severe heart disease, etc.)
* Difficulties in understanding and speaking Danish (eg. due to dementia)
* Place of residence outside Gentofte Hospital admission area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Composite outcome of 1 year mortality or hospital readmission | 12 months
  It is all cause mortality in 12 months follow-up period.. Readmission is the proportion of patients with at least 1 hospital readmission in 12 months follow-up period. Intention-to-treat analysis.Secondarily per-protocol analysis.

SECONDARY OUTCOMES:
All cause mortality and time to death | 12 months
All cause hospital readmission and time to readmission | 12 months
  Proportion of patients with at least 1 hospital readmission of any cause
Hospital readmission by respiratory cause | 12 months
Health related quality of life | 6 months
  Measured by COPD Assessment TEST (CAT)
Dyspnea | 6 months
  Measured by Medical Respiratory Council (MRC) dyspnea scale
Exercise performance | 6 months
  Composite measure by Incremental Shuttle Walk Test (ISWT) and Endurance Shuttle Walk Test (ESWT)

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Respiratory medicine, UH Gentofte, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No